CLINICAL TRIAL: NCT06477458
Title: Application of Deep Learning in CT Imaging of Elective Thoracic Surgery Patients: Assessing Preoperative Abnormal Pulmonary Function
Brief Title: Deep Learning for Preoperative Pulmonary Assessment in Thoracic CT
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Jianxing He, Director, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: ES-2024-091-02
Record Dates: First submitted 2024-06-21; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Elective Thoracic Surgery; Pulmonary Function; Deep Learning

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Single inspiratory phase cohort: Patients in this cohort undergo single inspiratory phase CT and pulmonary function tests preoperatively.
  Interventions: Other: Single inspiratory phase computed tomography.
- Respiratory dual-phase cohort: Patients in this cohort undergo respiratory dual-phase CT and pulmonary function tests preoperatively.
  Interventions: Other: Respiratory dual-phase computed tomography.

INTERVENTIONS:
Other: Single inspiratory phase computed tomography. — Utilizing deep learning technology in conjunction with single inspiratory phase computed tomography images to accurately predict the pulmonary function indicators of preoperative thoracic surgery patients.
  Groups: Single inspiratory phase cohort
Other: Respiratory dual-phase computed tomography. — Utilizing deep learning technology in conjunction with respiratory dual-phase computed tomography images to accurately predict the pulmonary function indicators of preoperative thoracic surgery patients.
  Groups: Respiratory dual-phase cohort

SUMMARY:
The trial was designed as a single-centre, non-interventional prospective observational study to utilize deep learning technology combined with computed tomography (CT) images to precisely predict the pulmonary function indicators of thoracic surgery preoperative patients.

DETAILED DESCRIPTION:
Preoperative pulmonary function tests are crucial in assessing perioperative complications or mortality risks and providing decision support for thoracic surgery. However, traditional pulmonary function assessment methods have significant limitations, including long testing durations, difficulties in patient cooperation, high false-negative rates, and numerous contraindications. Thus, our study optimized the final model based on 1500 single inspiratory phase CTs by transferring model parameters trained on 500 dual-phase respiratory CTs, enhancing its predictive capabilities for pulmonary function. This adjustment suits real-world application demands, offering more convenient, comprehensive, and personalized preoperative pulmonary function assessment support. Our study optimized the final model based on 1500 single inspiratory phase CTs by transferring model parameters trained on 500 dual-phase respiratory CTs, enhancing its predictive capabilities for pulmonary function. This adjustment suits real-world application demands, offering more convenient, comprehensive, and personalized preoperative pulmonary function assessment support.

ELIGIBILITY:
Inclusion Criteria:

* (1) Signing of the informed consent form;
* (2) Male or female, aged 18-75 years;
* (3) Undergoing elective thoracic surgery;
* (4) Good preoperative pulmonary function cooperation and complete reporting;
* (5) Preoperative chest single/dual phase CT scans without significant artefacts and with complete imaging;
* (6) The interval between preoperative pulmonary function and single/dual phase CT scans does not exceed one month.

Exclusion Criteria:

* (1) Poor preoperative pulmonary function cooperation or missing reports;
* (2) Preoperative chest single/dual phase CT scans exhibit significant artefacts or image omission;
* (3) The interval between preoperative pulmonary function and single/dual phase CT scans exceeds one month;
* (4) Complication with severe respiratory disorders (such as lung transplantation, pneumothorax, giant bullae, etc.);
* (5) Coexisting with other severe functional impairments;
* (6) Patients with obstructive lesions such as airway or esophageal stenosis;
* (7) Height beyond the predicted equation range (Female < 1.45m; Male < 1.55m);
* (8) Medication use before pulmonary function testing that does not meet the cessation guidelines;
* (9) Pulmonary function report quality graded D-F.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective Thoracic Surgery Patients
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Mean Absolute Error（MAE） | 2 years
  Used to assess the discrepancy between pulmonary function predictions made by the deep learning algorithm and actual results obtained from pulmonary function tests (measured with a spirometer).

SECONDARY OUTCOMES:
Concordance Correlation Coefficient（CCC） | 2 years
  Used to assess the discrepancy between pulmonary function predictions made by the deep learning algorithm and actual results obtained from pulmonary function tests (measured with a spirometer).

CONTACTS AND LOCATIONS:
Overall Officials: Jianxing He, MD, Principal Investigator — Department of Cardiothoracic Surgery, the First Affiliated Hospital of Guangzhou Medical College
Locations (1):
- Department of Cardiothoracic Surgery, the First Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong, China